CLINICAL TRIAL: NCT01409616
Title: A Randomized, Open-label, Two-period Crossover Study in Healthy Male Subjects to Evaluate the Pharmacodynamic Effect of Darexaban (YM150) on Acetyl Salicylic Acid (ASA) and of Darexaban on the Combination of ASA and Clopidogrel at Steady State
Brief Title: To Evaluate Whether Acetyl Salicylic Acid (Aspirin), the Combination of Aspirin and Clopidogrel and Darexaban (YM150) Interact in Their Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 150-CL-035; 2007-007036-26 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-04 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2011-08

CONDITIONS: Pharmacodynamic Interaction; Healthy Subjects
Keywords: Pharmacodynamics; darexaban; Acetyl Salicylic Acid; clopidogrel; YM150; Phase 1
MeSH Terms: interventions — darexaban; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment arm A (Experimental): ASA, wash-out (w.o.), ASA + darexaban
  Interventions: Drug: darexaban; Drug: Acetyl Salicylic Acid
- Treatment arm B (Experimental): ASA + darexaban, w.o., ASA
  Interventions: Drug: darexaban; Drug: Acetyl Salicylic Acid
- Treatment arm C (Experimental): ASA, w.o., darexaban (double dose) + ASA
  Interventions: Drug: darexaban (double dose); Drug: Acetyl Salicylic Acid
- Treatment arm D (Experimental): darexaban (double dose) + ASA, w.o., ASA
  Interventions: Drug: darexaban (double dose); Drug: Acetyl Salicylic Acid
- Treatment arm E (Experimental): ASA + clopidogrel, w.o., ASA + clopidogrel + darexaban
  Interventions: Drug: darexaban; Drug: Acetyl Salicylic Acid; Drug: clopidogrel
- Treatment arm F (Experimental): ASA + clopidogrel + darexaban, w.o., ASA + clopidogrel
  Interventions: Drug: darexaban; Drug: Acetyl Salicylic Acid; Drug: clopidogrel
- Treatment arm G (Experimental): ASA + clopidogrel, w.o., darexaban (double dose) + ASA + clopidogrel
  Interventions: Drug: darexaban (double dose); Drug: Acetyl Salicylic Acid; Drug: clopidogrel
- Treatment arm H (Experimental): darexaban (double dose) + ASA + clopidogrel, w.o., ASA + clopidogrel
  Interventions: Drug: darexaban (double dose); Drug: Acetyl Salicylic Acid; Drug: clopidogrel

INTERVENTIONS:
Drug: darexaban — oral
  Other Names: YM150
  Arms: Treatment arm A; Treatment arm B; Treatment arm E; Treatment arm F
Drug: darexaban (double dose) — oral
  Other Names: YM150
  Arms: Treatment arm C; Treatment arm D; Treatment arm G; Treatment arm H
Drug: Acetyl Salicylic Acid — oral
  Other Names: Aspirin
Drug: clopidogrel — oral
  Other Names: Plavix
  Arms: Treatment arm E; Treatment arm F; Treatment arm G; Treatment arm H

SUMMARY:
The primary objective of this study is to evaluate whether ASA, the combination of ASA and clopidogrel, and darexaban, which have different effects on blood coagulation, influence each other in their effects. Also it will be investigated whether the blood levels of either drug are influenced by the presence of the other drug. In addition, the safety and tolerability of each drug and the combination of the drugs will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5-30.0 kg/m2
* Male subjects must be non-fertile, i.e. surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies

Exclusion Criteria:

* Known or suspected hypersensitivity to darexaban or ASA or any components of the formulation used
* Any of the liver function tests (i.e. ALT, AST and bilirubin) above the upper limit of normal at repeated measures
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampicin) in the 3 months prior to admission to the Clinical Unit.
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse, or smoking of more than 10 cigarettes (or equivalent) or more than 21 units (210 g) of alcohol per week within the 3 months prior to study
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacodynamics of darexaban | Baseline and up to 24 hours after six days of dosing of darexaban, ASA, clopidogrel, or a combination

SECONDARY OUTCOMES:
Assessment of pharmacodynamics of ASA and a combination of ASA and clopidogrel | Baseline and up to 24 hours after six days of dosing of darexaban, ASA, clopidogrel, or a combination
Pharmacokinetics of ASA and the combination of ASA and clopidogrel assessed by plasma concentration | Plasma samples are taken until 24 hours after six days of dosing of ASA, a combination of ASA and clopidogrel, or the combination with darexaban
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | 6 days for each of the 2 treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.; Principal Investigator, Principal Investigator — SGS Aster, Paris, France
Locations (1):
- SGS Aster, Paris, France